CLINICAL TRIAL: NCT04098224
Title: Nutrition Monitoring and Feeding Optimization With the smART+ System
Brief Title: Nutrition Monitoring and Feeding Optimization With the smART+ System - Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ART Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CRO-C-2822
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Aspiration Pneumonia; Malnutrition
MeSH Terms: conditions — Pneumonia, Aspiration; Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Device - Treated (Experimental): Subjects connected to the investigational device smART+
  Interventions: Device: smART+ System
- Control Group (No Intervention): treated according to local Standard of Care.

INTERVENTIONS:
Device: smART+ System — Utilizing the smART+ System to provide feeding optimization to the patient
  Arms: Interventional Device - Treated

SUMMARY:
The smART+ is a comprehensive modular patient care system intended for ICU patients.

The main purpose of the study is the optimization of the delivery of nutrition.

The use of the smART+ Feeding tube includes a feature of facilitating correct tube placement and alerting when the tube is displaced during ongoing use. The system will automatically stop feeding if displacement is detected. If a massive reflux episode is detected by the system, a balloon located on the tube will automatically inflate and automatic GRV (Gastric Residual Volume) feature will open to prevent gastric content from regurgitating to the esophagus.

In addition to tube placement, the system allows to obtain REE (Resting Energy Expenditure) measurements and calculates the optimized nutritional values required by the patient. Furthermore, the system optimizes feeding by compensating for any lost feeding time or discarded nutritional content that was discarded via the GRV (Gastric Residual Volume).

Study participants will be randomly assigned to a study group:

Group A- ICU patients receiving the investigational device ("Treated"). Group B- Control group.

DETAILED DESCRIPTION:
Mechanically ventilated patients are unable to take food orally and therefore are dependent on enteral nutrition for provision of both energy and protein requirements. The conditions of ICU patients dramatically change throughout their ICU stay; "diseases, like particularly sepsis, trauma and burns, cause clinically relevant increase in resting energy expenditure (REE) of between 40% - 80%," and most patients do not reach their required protein and caloric targets. The American association for Parenteral and Enteral Nutrition (ASPEN) recommends that for patients who are at high risk for malnutrition, efforts should be made to provide >80% of the estimated or calculated energy and protein goal within 48-72 hours, starting with half the patient's calorie goal with the rate slowly increasing over time, in order to achieve the clinical benefit of enteral nutrition over the first week of hospitalization. However, studies have shown that more than 74% of ICU patients failed to receive at least 80% of their prescribed nutrition.

Predictive equations (such as Harris-Benedict equation) or a simple weight-based formula (48.1% and 48.7% respectively) have therefore been the most practiced methods of determining energy needs; however, the literature clearly indicates that each equation has a large potential for error. This makes it difficult to accurately predict an individual patient's energy requirements during critical illness. In general, predictive equations estimate accurately only 50% of the time in ICU patients, leading to over or under evaluation of the nutritional needs and inducing over or underfeeding. Numerous meta-analyses have demonstrated the poor value of predictive equations variability that is increased because body weight remains a value difficult to accurately assess.

To overcome the inaccuracy in determining the patient's energy consumption and the accompanying problems, the European Society for Parenteral and Enteral Nutrition (ESPEN) guidelines recommend to determine patients' REE based on indirect calorimetry or VCO2-based equation (VCO2 x 8.19). Unfortunately, this is not performed continuously during the course of enteral feeding to assess the ever-changing nutritional needs of the patient. Estimations showed that only 2% of ICUs were regularly using REE / indirect calorimetry,11 and therefore they must resort to performing a one-time calculation of the patient's energy consumption to manually calculate the caloric intake, food type and feeding rate.

This study aims to assess the accuracy of the smART+ System's REE module, compared to (1) the FDA-cleared COSMED device, and (2) nutritional calculations conducted with predictive equations regularly used by the clinical staff at the site.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years or older
* Patient that have already been admitted to the ICU (no more than 48 hours before enrollment)
* Expected to be ventilated at least 48 hours after enrollments.
* Patient requires enteral feeding (by naso/oro-gastric feeding tube)

Exclusion Criteria:

* Pregnant women
* Known anatomical anomalies of the nose, oral cavity esophagus or the stomach that may prevent/hinder the ability to insert the feeding tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Kagan, MD, Principal Investigator — Beilinson Hospital
Locations (1):
- Beilinson Hospital, Petah Tikva, Isreal, Israel

REFERENCES:
- [Derived] Kagan I, Hellerman-Itzhaki M, Bendavid I, Statlender L, Fishman G, Wischmeyer PE, de Waele E, Singer P. Controlled enteral nutrition in critical care patients - A randomized clinical trial of a novel management system. Clin Nutr. 2023 Sep;42(9):1602-1609. doi: 10.1016/j.clnu.2023.06.018. Epub 2023 Jul 7. PMID 37480797

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interventional Device - Treated | Control Group
Started | 50 | 50
Completed | 45 | 47
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Patient not required enteral feeding | 1 | 0
Not completed — Patient failure nasogastric tube | 1 | 0
Not completed — Patient early extubation | 1 | 3

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional Device - Treated | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (17.5) | 62.1 (16.0) | 60.7 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 39 | 34 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 50 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 50 | 50 | 100
BMI body mass index [Mean (Standard Deviation); unit: KG/M^2] | 29.2 (7.3) | 29.5 (8.8) | 29.3 (8.1)
APACHE II Acute Physiology and Chronic Healthy Evaluation II [Mean (Standard Deviation); unit: units on a scale] — APACHE II is a severity-of-disease classification system. It is applied within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
  units on a scale | 22.4 (6.9) | 22.3 (7.0) | 22.4 (6.9)
Time to Intensive Care Unit administration [Mean (Standard Deviation); unit: Hours] | 24.5 (11.7) | 28.3 (11.4) | 26.4 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Nutrition Optimization
Description: Optimization of the delivery of nutrition by the smART+ System as compared to standard of care, by automatically calculating and administering enteral feeding better than standard of care (REE or Calorimeter).
  The primary endpoint was the average feeding deviation between Days 2-14. Feeding deviation percentage was defined as the percentage of deviation from the nutrition target, calculated as the absolute value of 100 X (volume of nutrition delivered (mL) / the volume intended to be delivered (VTBD; mL))
Time Frame: 2 days-14 days
Measure: Mean (Standard Deviation); unit: percentage of feeding efficiency
Arm/Group | Interventional Device - Treated | Control Group
Number analyzed (Participants) | 48 | 50
percentage of feeding efficiency | 89.5 (13.0) | 65 (18.0)

2. Secondary Outcome: Device Safety According to Occurrence or Absence of Related AE Adverse Event or SAE Serious Adverse Events
Description: Safe use of the entire system will be assessed based on the occurrence of device-related AE adverse event or SAE Serious Adverse Events.
Time Frame: 2 days-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Device - Treated | Control Group
Number analyzed (Participants) | 50 | 50
Participants
  Adverse event related to device | 0 | 0
  Death not related to device | 3 | 3

3. Secondary Outcome: Decrease in Intensive Critical Unit Length of Stay
Description: Measured from admission to Intensive Critical Unit until the decision to discharge is ordered.
Time Frame: from admission to discharge from ICU ('ICU length of stay')
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Interventional Device - Treated | Control Group
Number analyzed (Participants) | 50 | 50
Days | 10.37 (7.01) | 13.65 (9.16)

4. Secondary Outcome: Reduction of Number of Patients With VAE (Ventilation Associated Events)
Description: Ventilated associated events (VAE) was evaluated by modifications of FIO2 fraction of inspired oxygen (above .2) or PEEP Positive end-expiratory pressure (above 3 cm H20) requirements that were longer than 48 hours [per the CDC Centers for Disease Control and Prevention definition and clinical judgment of the interpreting physician]
Time Frame: 2 days-14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Device - Treated | Control Group
Number analyzed (Participants) | 50 | 50
Participants | 1 | 5

5. Secondary Outcome: Decrease in ICU Ventilation Days
Description: Evaluated by the number of hours of End-tidal CO2 from the hospital electronic records
Time Frame: from admission to discharge from ICU ('ICU length of stay') up to 14 days.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Interventional Device - Treated | Control Group
Number analyzed (Participants) | 50 | 50
Days | 9.52 (7.32) | 12.78 (8.74)

6. Secondary Outcome: Decrease in Workload Related to Nurse Gastric Residual Volume (GRV) Time
Description: The change in workload could be estimated by using the estimated nursing time that was expended for GRV activities, and the amounts of GRV removed from the patient obtained through the hospital's electronic records.
Time Frame: 2 days-14 days
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/day
Arm/Group | Interventional Device - Treated | Control Group
Number analyzed (Participants) | 50 | 50
ml/day
  Daily total amount of GRV [ml/day] | 124.25 [100.03 to 148.46] | 166.10 [145.93 to 186.27]
  Max GRV per event in one day [ml/d] | 33.3941 [18.8106 to 47.9777] | 114.95 [102.82 to 127.08]

7. Secondary Outcome: Assessment of Urine Flow Monitoring Related to Patient Condition
Description: Patient lab results obtained through the hospital's electronic records will be analyzed against smART+ system urine alerts to determine if the alerts will be useful in the diagnosis
Time Frame: 2 days-14 days
Population: In order to assess this endpoint a larger sample size is required. This secondary endpoint was omitted from the study because the study enrollment was stopped after the primary endpoint of feeding efficiency was achieved (100 patients enrolled).
Arm/Group | Interventional Device - Treated | Control Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Convenience of Use of the System and the User Interface (by Subjective Staff Questionnaire)
Description: Subjective staff questionnaire to be completed by all personnel involved in the study, to assess usability. In order to assess this endpoint a larger sample size is required. This secondary endpoint was omitted from the study because the study enrollment was stopped after the primary endpoint of feeding efficוency was achieved (100 patients enrolled).
Time Frame: Throughout the study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse event for each patient was collected form the day of screening visit until the day of completing the study , totally 14 days .
Arm/Group | Interventional Device - Treated | Control Group
All-Cause Mortality (participants affected / at risk) | 3/50 | 3/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 3/50
Other Adverse Events (participants affected / at risk) | 35/50 | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional Device - Treated (N=50) | Control Group (N=50)
Post COVID 19 (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Desaturation (Cardiac disorders) | 0 | 1
Respiratory and hemodynamic deterioration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Septic shock deterioration (Infections and infestations) | 1 | 0
Severe progressive hypoxemic and hemodynamic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional Device - Treated (N=50) | Control Group (N=50)
New infection in blood (Infections and infestations) | 9 | 11
New infection in sputum (Infections and infestations) | 20 | 23
New infection in broncial lavage (Infections and infestations) | 2 | 7
Atrial fibralation (Cardiac disorders) | 2 | 4
Bradycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 3
Low hemoglobin level (Blood and lymphatic system disorders) | 2 | 3
Self nasogastric tube removal (Product Issues) | 3 | 0
Hypomagnesemia (General disorders) | 0 | 1
Fever (General disorders) | 1 | 2
Pressure sores (General disorders) | 0 | 1
High blood pressure (General disorders) | 0 | 2
Lower blood pressure (General disorders) | 1 | 0
Hypophosphatemia (General disorders) | 2 | 2
Massive diarrhea (Metabolism and nutrition disorders) | 0 | 1
High GRV (Metabolism and nutrition disorders) | 1 | 0
Respiratory rate deterioration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary infiltate (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Left atelectasis (Ear and labyrinth disorders) | 0 | 1
Tonic clonic seizure (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was designed to detect an effect size of 0.45 for 100 patients per group (200 total enrollment) using a two- group test with a 0.05 two-sided signiﬁcance level. A single interim analysis was planned after 100 patients. The trial was stopped after the interim analysis of the available data of the 100 enrolled patients, as sufficient data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04098224/Prot_SAP_000.pdf